CLINICAL TRIAL: NCT01162421
Title: Radiographic, Clinical and Patient Outcomes in a Multicenter, Open Label Phase IV Randomized Trial of Earlier Adalimumab Introduction Therapy Versus Later Introduction as Per Standard of Care After Initial Methotrexate Failure in Early Rheumatoid Arthritis Patients
Brief Title: A Canadian Study to Evaluate Early Use of Adalimumab After Methotrexate Failure in Early Rheumatoid Arthritis
Acronym: RADAR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Collaborators: Mount Sinai Hospital, Canada (Other)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: W12-122
Record Dates: First submitted 2010-05-25; First posted 2010-07-14 (Estimated); Results first posted 2016-11-01 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-09

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; Anti-Inflammatory; Biological Therapy; adalimumab; Disease-Modifying Antirheumatic Drugs; Antirheumatic Agents; Agents
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Adalimumab; Methotrexate

ARMS (2):
- Early Adalimumab (Experimental): Participants in the Early Adalimumab arm will receive adalimumab and methotrexate at Baseline and every other week for study duration.
  Interventions: Biological: adalimumab; Drug: Methotrexate
- Standard of Care (Active Comparator): Participants in the Standard of Care arm will receive methotrexate and other disease modifying antirheumatic drugs as per local treatment guidelines and study doctor's judgement. Adalimumab may be initiated after a minimum of 6 months.
  Interventions: Biological: adalimumab; Drug: Methotrexate

INTERVENTIONS:
Biological: adalimumab — Study drug will be provided to participants in Early Adalimumab arm as a sterile, preservative-free solution for subcutaneous injection, contained in a pre-filled syringe housed in a pen device (pre-filled pen). 40 mg of adalimumab will be administered subcutaneously at Baseline and then every other week for 24 months. Adalimumab may be initiated in participants in standard of care (SOC) arm after a minimum of 6 months of treatment recommended by their study doctor.
  Other Names: ABT-D2E7; Humira
Drug: Methotrexate — Participants in both arms will receive a methotrexate regimen based on local guidelines and their study doctor's judgment.
  Other Names: Trexall; Rheumatrex

SUMMARY:
A Canadian study to evaluate early use of adalimumab after methotrexate failure in early rheumatoid arthritis. The study hypothesis will verify if adalimumab effectively reduces joint damage in more participants when introduced earlier than in current practice.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has a diagnosis of Rheumatoid Arthritis as defined by the 1987-revised American College of Rheumatology-classification criteria and has disease duration of less than 2 years from diagnosis.
2. Subject must have been on a dose of methotrexate therapy either subcutaneously or orally administered (15-25 mg/week) for at least 3 months prior to baseline visit and has had an inadequate response to treatment defined as having a Disease Activity Score DAS28 > 3.2 (at Screening visit).
3. Subject must also meet the following three criteria (at screening visit): at least 4 swollen joints out of 66 assessed; at least 4 tender joints out of 68 assessed; subject must have an elevated erythrocyte sedimentation rate >/= 20 mm/1h or C-reactive protein > upper limit of normal.
4. Subject must fulfill at least one of the following three criteria: history of rheumatoid factor positive; history of at least one erosion on X-ray or magnetic resonance imaging; history of anti-cyclic-citrullinated protein antibody positive.

Exclusion Criteria:

1. Subject has previous exposure to any biologic therapy including adalimumab.
2. Prior disease-modifying antirheumatic drugs triple therapy with methotrexate.
3. Subject has been treated with intra-articular or parenteral administration of corticosteroids in the preceding 4 weeks prior to baseline visit. Inhaled corticosteroids for stable medical conditions are allowed.
4. Subject has undergone joint surgery within the preceding two months (at joints to be assessed within the study) of Baseline.
5. Subject has a poorly controlled medical condition, such as uncontrolled diabetes, unstable heart disease, congestive heart failure, recent cerebrovascular accidents and any other condition which, in the opinion of the Investigator, would put the subject at risk by participating in the study.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2010-09; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christina Pelizon, MD, Study Director — AbbVie Corporation

REFERENCES:
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard of Care: Participants received methotrexate and other disease modifying antirheumatic drugs as per local treatment guidelines and study doctor's judgement. Adalimumab may have been initiated after a minimum of 6 months.
- Early Adalimumab: Participants received 40 mg of adalimumab administered subcutaneously at Baseline and then every other week for 24 months. Participants received a methotrexate regimen based on local guidelines and their study doctor's judgment.
Period: Overall Study
Arm/Group | Standard of Care | Early Adalimumab
Started | 37 | 40
Completed | 29 | 27
Not Completed | 8 | 13
Not completed — Did not receive study drug | 2 | 1
Not completed — Adverse Event | 2 | 5
Not completed — Lost to Follow-up | 0 | 2
Not completed — Lack of Efficacy | 2 | 2
Not completed — Other | 2 | 3

BASELINE CHARACTERISTICS:
Population: Intent-to-treat population: all participants who were randomized and received at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care | Early Adalimumab | Total
Number analyzed (Participants) | 35 | 39 | 74
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.8 (10.46) | 51.9 (11.55) | 52.8 (11.01)
Age, Customized [Number; unit: participants]
  < 65 years | 30 | 34 | 64
  >/= 65 years | 5 | 5 | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 26 | 50
  Male | 11 | 13 | 24

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With No Radiographic Progression at Month 12
Description: Radiographic progression was defined as change from Baseline in the modified Total Sharp Score (mTSS) of ≤ 0.5 units). The mTSS is a measure of change in joint health: digitized images of radiographs of hands and feet obtained at Screening and Month 12 were scored in a blinded manner. Joints were scored for erosions on a scale from 0 (no damage) to 5 (complete collapse) and joint space narrowing on a scale from 0 (no damage) to 4 (ankylosis or complete dislocation). Erosion scores and narrowing scores were added to obtain the mTSS (range = 0 [normal] to 398 [maximal disease]). An increase in mTSS from Baseline represents disease progression and/or joint worsening, no change represents halting of disease progression, and a decrease represents improvement.
Time Frame: Baseline, Month 12
Population: Intent-to-treat population: all participants who were randomized and received at least one dose of study drug. Last observation carried forward (LOCF): missing responses were imputed by carrying forward the last non-missing post-baseline observation.
Measure: Number; unit: percentage of participants
Arm/Group | Standard of Care | Early Adalimumab
Number analyzed (Participants) | 35 | 39
percentage of participants | 62.9 | 61.5
Statistical Analysis 1: Comparison: Standard of Care vs Early Adalimumab; Test type: Superiority or Other; p = 0.907, Chi-squared; P-value is based on two-sided Pearson's chi-square test; Difference in percentage = -1.3, 95% CI 2-sided [-23.4 to 20.8]

2. Secondary Outcome: Percentage of Participants With No Radiographic Progression at Month 6 and Month 24
Description: as for outcome 1
Time Frame: Baseline, Month 6, Month 24
Population: Intent-to-treat population: all participants who were randomized and received at least one dose of study drug (nonresponder imputation).
Measure: Number; unit: percentage of participants
Arm/Group | Standard of Care | Early Adalimumab
Number analyzed (Participants) | 35 | 39
percentage of participants
  Month 6 | 68.6 | 71.8
  Month 24 | 51.4 | 46.2
Statistical Analysis 1: Comparison: Standard of Care vs Early Adalimumab; Month 6; Test type: Superiority or Other; p = 0.762, Chi-squared; P-value is based on two-sided Pearson's chi-square test; Difference in percentage = 3.2, 95% CI 2-sided [-17.7 to 24.1]
Statistical Analysis 2: Comparison: Standard of Care vs Early Adalimumab; Month 24; Test type: Superiority or Other; p = 0.650, Chi-squared; P-value is based on two-sided Pearson's chi-square test; Difference in percentage = -5.3, 95% CI 2-sided [-28.1 to 17.5]

3. Secondary Outcome: Change From Baseline in mTSS at Months 6, 12 and 24
Description: The mTSS is a measure of change in joint health: digitized images of radiographs of hands and feet obtained at Screening and Month 12 were scored in a blinded manner. Joints were scored for erosions on a scale from 0 (no damage) to 5 (complete collapse) and joint space narrowing on a scale from 0 (no damage) to 4 (ankylosis or complete dislocation). Erosion scores and narrowing scores were added to obtain the mTSS (range = 0 [normal] to 398 [maximal disease]). An increase in mTSS from Baseline represents disease progression and/or joint worsening, no change represents halting of disease progression, and a decrease represents improvement.
Time Frame: Baseline, Month 6, Month 12, Month 24
Population: Intent-to-treat population: all participants who were randomized and received at least one dose of study drug; n=number of participants with an assessment at Baseline and given timepoint (observed cases).
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Standard of Care | Early Adalimumab
Number analyzed (Participants) | 35 | 39
units on a scale
  Month 6; n=34, 36 | 0.88 (0.273) | 0.02 (0.266)
  Month 12; n=30, 34 | 1.62 (0.486) | 0.16 (0.457)
  Month 24; n=28, 21 | 2.24 (0.912) | 0.01 (1.055)
Statistical Analysis 1: Comparison: Standard of Care vs Early Adalimumab; Month 6; Test type: Superiority or Other; p = 0.027, ANCOVA — P-values are two-sided and are based on repeated measures ANCOVA model with treatment group and visit as the fixed effects and baseline value as the covariate; The a priori threshold for statistical significance is P= 0.05; Least squares (LS) Mean Difference = -0.86, 95% CI 2-sided [-1.62 to -0.10], Standard Error of Mean 0.382
Statistical Analysis 2: Comparison: Standard of Care vs Early Adalimumab; Month 12; Test type: Superiority or Other; p = 0.033, ANCOVA — [p-value comment as in outcome 3, analysis 1]; The a priori threshold for statistical significance is P= 0.05; LS Mean Difference = -1.46, 95% CI 2-sided [-2.79 to -0.12], Standard Error of Mean 0.667
Statistical Analysis 3: Comparison: Standard of Care vs Early Adalimumab; Month 24; Test type: Superiority or Other; p = 0.120, ANCOVA — [p-value comment as in outcome 3, analysis 1]; LS Mean Difference = -2.22, 95% CI 2-sided [-5.05 to 0.60], Standard Error of Mean 1.403

4. Secondary Outcome: Percentage of Participants With Rapid Radiographic Progression at Month 12
Description: Radiographic progression was defined as a change from Baseline in mTSS that is ≥ 5 units. The mTSS is a measure of change in joint health: digitized images of radiographs of hands and feet obtained at Screening and Month 12 were scored in a blinded manner. Joints were scored for erosions on a scale from 0 (no damage) to 5 (complete collapse) and joint space narrowing on a scale from 0 (no damage) to 4 (ankylosis or complete dislocation). Erosion scores and narrowing scores were added to obtain the mTSS (range = 0 [normal] to 398 [maximal disease]). An increase in mTSS from Baseline represents disease progression and/or joint worsening, no change represents halting of disease progression, and a decrease represents improvement.
Time Frame: Month 12
Population: Intent-to-treat population: all participants who were randomized and received at least one dose of study drug ith an assessment (nonresponder imputation).
Measure: Number; unit: percentage of participants
Arm/Group | Standard of Care | Early Adalimumab
Number analyzed (Participants) | 34 | 39
percentage of participants | 14.3 | 2.6
Statistical Analysis 1: Comparison: Standard of Care vs Early Adalimumab; Test type: Superiority or Other; p = 0.095, Fisher Exact — P-value is based on two sided Fisher's exact test; Difference in percentage = -11.7, 95% CI 2-sided [-27.0 to 1.6] — Confidence interval is based on Wilson confidence limits

5. Secondary Outcome: Percentage of Participants With American College of Rheumatology 20% (ACR20) Response at Months 3, 6, 9, 12, 18 and 24
Description: A participant is an ACR20 responder if the following 3 criteria for improvement from Baseline are met:
  * ≥ 20% improvement in tender joint count;
  * ≥ 20% improvement in swollen joint count; and
  * ≥ 20% improvement in at least 3 of the 5 following parameters: -
    * Physician global assessment of disease activity
    * Patient global assessment of disease activity
    * Patient assessment of pain
    * Disability Index of the Health Assessment Questionnaire
    * Acute phase reactant (erythrocyte sedimentation rate/C-reactive protein [CRP]).
Time Frame: Baseline, Months 3, 6, 9, 12, 18, 24
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Standard of Care | Early Adalimumab
Number analyzed (Participants) | 35 | 39
percentage of participants
  Month 3 | 57.1 | 69.2
  Month 6 | 37.1 | 64.1
  Month 9 | 60.0 | 66.7
  Month 12 | 68.6 | 56.4
  Month 18 | 65.7 | 51.3
  Month 24 | 65.7 | 46.2
Statistical Analysis 1: Comparison: Standard of Care vs Early Adalimumab; Month 3; Test type: Superiority or Other; p = 0.281, Chi-squared; P-value is based on two-sided Pearson's chi-square test; Difference in percentage = 12.1, 95% CI 2-sided [-9.79 to 33.97]
Statistical Analysis 2: Comparison: Standard of Care vs Early Adalimumab; Month 6; Test type: Superiority or Other; p = 0.021, Chi-squared — The a priori threshold for statistical significance is P=0.05; P-value is based on two-sided Pearson's chi-square test; Difference in percentage = 27.0, 95% CI 2-sided [4.98 to 48.93]
Statistical Analysis 3: Comparison: Standard of Care vs Early Adalimumab; Month 9; Test type: Superiority or Other; p = 0.552, Chi-squared; P-value is based on two-sided Pearson's chi-square test; Difference in percentage = 6.7, 95% CI 2-sided [-15.29 to 28.63]
Statistical Analysis 4: Comparison: Standard of Care vs Early Adalimumab; Month 12; Test type: Superiority or Other; p = 0.281, Chi-squared; P-value is based on two-sided Pearson's chi-square test; Difference in percentage = -12.2, 95% CI 2-sided [-34.04 to 9.72]
Statistical Analysis 5: Comparison: Standard of Care vs Early Adalimumab; Month 18; Test type: Superiority or Other; p = 0.209, Chi-squared; P-value is based on two-sided Pearson's chi-square test; Difference in percentage = -14.4, 95% CI 2-sided [-36.64 to 7.78]
Statistical Analysis 6: Comparison: Standard of Care vs Early Adalimumab; Month 24; Test type: Superiority or Other; p = 0.091, Chi-squared; P-value is based on two-sided Pearson's chi-square test; Difference in percentage = -19.6, 95% CI 2-sided [-41.74 to 2.62]

6. Secondary Outcome: Percentage of Participants With American College of Rheumatology 50% (ACR50) Response at Months 3, 6, 9, 12, 18 and 24
Description: A participant is an ACR50 responder if the following 3 criteria for improvement from Baseline are met:
  * ≥ 50% improvement in tender joint count;
  * ≥ 50% improvement in swollen joint count; and
  * ≥ 50% improvement in at least 3 of the 5 following parameters:
    * Physician global assessment of disease activity
    * Patient global assessment of disease activity
    * Patient assessment of pain
    * Disability Index of the Health Assessment Questionnaire
    * Acute phase reactant (erythrocyte sedimentation rate/CRP).
Time Frame: Baseline, Months 3, 6, 9, 12, 18, 24
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Standard of Care | Early Adalimumab
Number analyzed (Participants) | 35 | 39
percentage of participants
  Month 3 | 22.9 | 38.5
  Month 6 | 22.9 | 43.6
  Month 9 | 40.0 | 48.7
  Month 12 | 34.3 | 43.6
  Month 18 | 45.7 | 38.5
  Month 24 | 42.9 | 33.3
Statistical Analysis 1: Comparison: Standard of Care vs Early Adalimumab; Month 3; Test type: Superiority or Other; p = 0.148, Chi-squared; P-value is based on two-sided Pearson's chi-square test; Difference in percentage = 15.6, 95% CI 2-sided [-5.05 to 36.26]
Statistical Analysis 2: Comparison: Standard of Care vs Early Adalimumab; Month 6; Test type: Superiority or Other; p = 0.060, Chi-squared; P-value is based on two-sided Pearson's chi-square test; Difference in percentage = 20.7, 95% CI 2-sided [-0.14 to 41.61]
Statistical Analysis 3: Comparison: Standard of Care vs Early Adalimumab; Month 9; Test type: Superiority or Other; p = 0.451, Chi-squared; P-value is based on two-sided Pearson's chi-square test; Difference in percentage = 8.7, 95% CI 2-sided [-13.85 to 31.29]
Statistical Analysis 4: Comparison: Standard of Care vs Early Adalimumab; Month 12; Test type: Superiority or Other; p = 0.413, Chi-squared; P-value is based on two-sided Pearson's chi-square test; Difference in percentage = 9.3, 95% CI 2-sided [-12.82 to 31.43]
Statistical Analysis 5: Comparison: Standard of Care vs Early Adalimumab; Month 18; Test type: Superiority or Other; p = 0.528, Chi-squared; P-value is based on two-sided Pearson's chi-square test; Difference in percentage = -7.3, 95% CI 2-sided [-29.74 to 15.23]
Statistical Analysis 6: Comparison: Standard of Care vs Early Adalimumab; Month 24; Test type: Superiority or Other; p = 0.399, Chi-squared; P-value is based on two-sided Pearson's chi-square test; Difference in percentage = -9.5, 95% CI 2-sided [-31.61 to 12.56]

7. Secondary Outcome: Percentage of Participants With American College of Rheumatology 70% (ACR70) Response at Months 3, 6, 9, 12, 18 and 24
Description: A participant is an ACR70 responder if the following 3 criteria for improvement from Baseline are met:
  * ≥ 70% improvement in tender joint count;
  * ≥ 70% improvement in swollen joint count; and
  * ≥ 70% improvement in at least 3 of the 5 following parameters: -
    * Physician global assessment of disease activity
    * Patient global assessment of disease activity
    * Patient assessment of pain
    * Disability Index of the Health Assessment Questionnaire
    * Acute phase reactant (erythrocyte sedimentation rate/CRP).
Time Frame: Months 3, 6, 9, 12, 18, 24
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Standard of Care | Early Adalimumab
Number analyzed (Participants) | 35 | 39
percentage of participants
  Month 3 | 2.9 | 15.4
  Month 6 | 8.6 | 28.2
  Month 9 | 22.9 | 25.6
  Month 12 | 14.3 | 30.8
  Month 18 | 20.0 | 30.8
  Month 24 | 40.0 | 23.1
Statistical Analysis 1: Comparison: Standard of Care vs Early Adalimumab; Month 3; Test type: Superiority or Other; p = 0.111, Fisher Exact; Difference in percentage = 12.5, 95% CI 2-sided [-1.70 to 27.06]
Statistical Analysis 2: Comparison: Standard of Care vs Early Adalimumab; Month 6; Test type: Superiority or Other; p = 0.031, Chi-squared — The a priori threshold for statistical significance is P=0.05; P-value is based on two-sided Pearson's chi-square test; Difference in percentage = 19.6, 95% CI 2-sided [2.74 to 36.53]
Statistical Analysis 3: Comparison: Standard of Care vs Early Adalimumab; Month 9; Test type: Superiority or Other; p = 0.780, Chi-squared; P-value is based on two-sided Pearson's chi-square test; Difference in percentage = 2.8, 95% CI 2-sided [-16.74 to 22.31]
Statistical Analysis 4: Comparison: Standard of Care vs Early Adalimumab; Month 12; Test type: Superiority or Other; p = 0.092, Chi-squared; P-value is based on two-sided Pearson's chi-square test; Difference in percentage = 16.5, 95% CI 2-sided [-2.07 to 35.04]
Statistical Analysis 5: Comparison: Standard of Care vs Early Adalimumab; Month 18; Test type: Superiority or Other; p = 0.290, Chi-squared; P-value is based on two-sided Pearson's chi-square test; Difference in percentage = 10.8, 95% CI 2-sided [-8.86 to 30.40]
Statistical Analysis 6: Comparison: Standard of Care vs Early Adalimumab; Month 24; Test type: Superiority or Other; p = 0.116, Chi-squared; P-value is based on two-sided Pearson's chi-square test; Difference in percentage = -16.9, 95% CI 2-sided [-37.86 to 4.01]

8. Secondary Outcome: Change From Baseline in Swollen Joint Count 66 at Months 3, 6, 9, 12, 18 and 24
Description: Sixty-six joints were assessed and classified as swollen/not swollen by pressure and joint manipulation on physical examination. The presence of swelling is scored 1 and no swelling is 0; range of score is 0-66, with higher scores indicating more swollen joints.
Time Frame: Baseline, Months 3, 6, 9, 12, 18, 24
Population: Intent-to-treat population: all participants who were randomized and received at least one dose of study drug with an assessment. LOCF: missing responses were imputed by carrying forward the last non-missing post-baseline observation.
Measure: Least Squares Mean (Standard Error); unit: swollen joints
Arm/Group | Standard of Care | Early Adalimumab
Number analyzed (Participants) | 35 | 38
swollen joints
  Month 3 | -5.6 (0.85) | -9.2 (0.81)
  Month 6 | -5.9 (0.81) | -10.4 (0.78)
  Month 9 | -8.1 (0.84) | -10.8 (0.80)
  Month 12 | -9.2 (0.69) | -11.3 (0.66)
  Month 18 | -9.4 (1.14) | -10.0 (1.09)
  Month 24 | -10.1 (0.83) | -10.6 (0.80)
Statistical Analysis 1: Comparison: Standard of Care vs Early Adalimumab; Month 3; Test type: Superiority or Other; p = 0.004, ANCOVA — [p-value comment as in outcome 3, analysis 1]; The a priori threshold for statistical significance is P=0.01; LS Mean Difference = -3.5, 95% CI 2-sided [-5.9 to -1.2], Standard Error of Mean 1.18
Statistical Analysis 2: Comparison: Standard of Care vs Early Adalimumab; Month 6; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; The a priori threshold for statistical significance is P=0.001; LS Mean Difference = -4.5, 95% CI 2-sided [-6.8 to -2.3], Standard Error of Mean 1.12
Statistical Analysis 3: Comparison: Standard of Care vs Early Adalimumab; Month 9; Test type: Superiority or Other; p = 0.021, ANCOVA — [p-value comment as in outcome 3, analysis 1]; The a priori threshold for statistical significance is P=0.05; LS Mean Difference = -2.7, 95% CI 2-sided [-5.1 to -0.4], Standard Error of Mean 1.16
Statistical Analysis 4: Comparison: Standard of Care vs Early Adalimumab; Month 12; Test type: Superiority or Other; p = 0.037, ANCOVA — [p-value comment as in outcome 3, analysis 1]; The a priori threshold for statistical significance is P=0.05; LS Mean Difference = -2.0, 95% CI 2-sided [-4.0 to -0.1], Standard Error of Mean 0.96
Statistical Analysis 5: Comparison: Standard of Care vs Early Adalimumab; Month 18; Test type: Superiority or Other; p = 0.702, ANCOVA — [p-value comment as in outcome 3, analysis 1]; LS Mean Difference = -0.6, 95% CI 2-sided [-3.7 to 2.5], Standard Error of Mean 1.58
Statistical Analysis 6: Comparison: Standard of Care vs Early Adalimumab; Month 24; Test type: Superiority or Other; p = 0.644, ANCOVA — [p-value comment as in outcome 3, analysis 1]; LS Mean Difference = -0.5, 95% CI 2-sided [-2.8 to 1.8], Standard Error of Mean 1.15

9. Secondary Outcome: Change From Baseline in Swollen Joint Count 28 at Months 3, 6, 9, 12, 18 and 24
Description: Twenty-eight joints were assessed and classified as swollen/not swollen by pressure and joint manipulation on physical examination. The presence of swelling is scored 1 and no swelling is 0; range of score is 0-28, with higher scores indicating more swollen joints.
Time Frame: Baseline, Months 3, 6, 9, 12, 18, 24
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: swollen joints
Arm/Group | Standard of Care | Early Adalimumab
Number analyzed (Participants) | 35 | 38
swollen joints
  Month 3 | -4.6 (0.64) | -6.5 (0.62)
  Month 6 | -4.5 (0.57) | -7.9 (0.55)
  Month 9 | -6.1 (0.58) | -8.3 (0.56)
  Month 12 | -6.9 (0.51) | -8.5 (0.49)
  Month 18 | -7.4 (0.68) | -8.1 (0.65)
  Month 24 | -7.6 (0.55) | -8.4 (0.53)
Statistical Analysis 1: Comparison: Standard of Care vs Early Adalimumab; Month 3; Test type: Superiority or Other; p = 0.039, ANCOVA — [p-value comment as in outcome 3, analysis 1]; The a priori threshold for statistical significance is P=0.05; LS Mean Difference = -1.9, 95% CI 2-sided [-3.7 to -0.1], Standard Error of Mean 0.89
Statistical Analysis 2: Comparison: Standard of Care vs Early Adalimumab; Month 6; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; The a priori threshold for statistical significance is P=0.001; LS Mean Difference = -3.4, 95% CI 2-sided [-5.0 to -1.8], Standard Error of Mean 0.79
Statistical Analysis 3: Comparison: Standard of Care vs Early Adalimumab; Month 9; Test type: Superiority or Other; p = 0.008, ANCOVA — [p-value comment as in outcome 3, analysis 1]; The a priori threshold for statistical significance is P=0.01; LS Mean Difference = -2.2, 95% CI 2-sided [-3.8 to -0.6], Standard Error of Mean 0.81
Statistical Analysis 4: Comparison: Standard of Care vs Early Adalimumab; Month 12; Test type: Superiority or Other; p = 0.028, ANCOVA — [p-value comment as in outcome 3, analysis 1]; The a priori threshold for statistical significance is P=0.05; LS Mean Difference = -1.6, 95% CI 2-sided [-3.0 to -0.2], Standard Error of Mean 0.71
Statistical Analysis 5: Comparison: Standard of Care vs Early Adalimumab; Month 18; Test type: Superiority or Other; p = 0.452, ANCOVA — [p-value comment as in outcome 3, analysis 1]; LS Mean Difference = -0.7, 95% CI 2-sided [-2.6 to 1.2], Standard Error of Mean 0.94
Statistical Analysis 6: Comparison: Standard of Care vs Early Adalimumab; Month 24; Test type: Superiority or Other; p = 0.343, ANCOVA — [p-value comment as in outcome 3, analysis 1]; LS Mean Difference = -0.7, 95% CI 2-sided [-2.3 to 0.8], Standard Error of Mean 0.77

10. Secondary Outcome: Change From Baseline in Tender Joint Count 68 at Months 3, 6, 9, 12, 18 and 24
Description: Sixty-eight joints were assessed and classified as tender/not tender by pressure and joint manipulation on physical examination. The presence of tenderness is scored 1 and no tenderness is 0; range of score is 0-68, with higher scores indicating more tender joints.
Time Frame: Baseline, Months 3, 6, 9, 12, 18, 24
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: tender joints
Arm/Group | Standard of Care | Early Adalimumab
Number analyzed (Participants) | 35 | 38
tender joints
  Month 3 | -9.3 (1.63) | -12.1 (1.56)
  Month 6 | -8.3 (1.38) | -15.5 (1.33)
  Month 9 | -11.2 (1.35) | -15.0 (1.30)
  Month 12 | -13.4 (1.41) | -14.1 (1.35)
  Month 18 | -13.4 (1.67) | -13.9 (1.60)
  Month 24 | -15.0 (1.32) | -15.8 (1.27)
Statistical Analysis 1: Comparison: Standard of Care vs Early Adalimumab; Month 3; Test type: Superiority or Other; p = 0.220, ANCOVA — [p-value comment as in outcome 3, analysis 1]; LS Mean Difference = -2.8, 95% CI 2-sided [-7.3 to 1.7], Standard Error of Mean 2.26
Statistical Analysis 2: Comparison: Standard of Care vs Early Adalimumab; Month 6; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; The a priori threshold for statistical significance is P=0.001; LS Mean Difference = -7.2, 95% CI 2-sided [-11.0 to -3.3], Standard Error of Mean 1.92
Statistical Analysis 3: Comparison: Standard of Care vs Early Adalimumab; Month 9; Test type: Superiority or Other; p = 0.050, ANCOVA — [p-value comment as in outcome 3, analysis 1]; The a priori threshold for statistical significance is P=0.05; LS Mean Difference = -3.7, 95% CI 2-sided [-7.5 to 0.0], Standard Error of Mean 1.87
Statistical Analysis 4: Comparison: Standard of Care vs Early Adalimumab; Month 12; Test type: Superiority or Other; p = 0.725, ANCOVA — [p-value comment as in outcome 3, analysis 1]; LS Mean Difference = -0.7, 95% CI 2-sided [-4.6 to 3.2], Standard Error of Mean 1.95
Statistical Analysis 5: Comparison: Standard of Care vs Early Adalimumab; Month 18; Test type: Superiority or Other; p = 0.837, ANCOVA — [p-value comment as in outcome 3, analysis 1]; LS Mean Difference = -0.5, 95% CI 2-sided [-5.1 to 4.1], Standard Error of Mean 2.31
Statistical Analysis 6: Comparison: Standard of Care vs Early Adalimumab; Month 24; Test type: Superiority or Other; p = 0.661, ANCOVA — [p-value comment as in outcome 3, analysis 1]; LS Mean Difference = -0.8, 95% CI 2-sided [-4.5 to 2.9], Standard Error of Mean 1.83

11. Secondary Outcome: Change From Baseline in Tender Joint Count 28 at Months 3, 6, 9, 12, 18 and 24
Description: Twenty-eight joints were assessed and classified as tender/not tender by pressure and joint manipulation on physical examination. The presence of tenderness is scored 1 and no tenderness is 0; range of score is 0-28, with higher scores indicating more tender joints.
Time Frame: Baseline, Months 3, 6, 9, 12, 18, 24
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: tender joints
Arm/Group | Standard of Care | Early Adalimumab
Number analyzed (Participants) | 35 | 38
tender joints
  Month 3 | -5.5 (0.93) | -7.4 (0.90)
  Month 6 | -5.7 (0.78) | -9.7 (0.74)
  Month 9 | -7.1 (0.86) | -9.6 (0.83)
  Month 12 | -8.4 (0.82) | -9.2 (0.79)
  Month 18 | -8.5 (0.94) | -9.1 (0.90)
  Month 24 | -9.4 (0.80) | -10.2 (0.77)
Statistical Analysis 1: Comparison: Standard of Care vs Early Adalimumab; Month 3; Test type: Superiority or Other; p = 0.156, ANCOVA — [p-value comment as in outcome 3, analysis 1]; LS Mean Difference = -1.9, 95% CI 2-sided [-4.4 to 0.7], Standard Error of Mean 1.29
Statistical Analysis 2: Comparison: Standard of Care vs Early Adalimumab; Month 6; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; The a priori threshold for statistical significance is P=0.001; LS Mean Difference = -4.0, 95% CI 2-sided [-6.1 to -1.9], Standard Error of Mean 1.08
Statistical Analysis 3: Comparison: Standard of Care vs Early Adalimumab; Month 9; Test type: Superiority or Other; p = 0.040, ANCOVA — [p-value comment as in outcome 3, analysis 1]; The a priori threshold for statistical significance is P=0.05; LS Mean Difference = -2.5, 95% CI 2-sided [-4.9 to -0.1], Standard Error of Mean 1.19
Statistical Analysis 4: Comparison: Standard of Care vs Early Adalimumab; Month 12; Test type: Superiority or Other; p = 0.492, ANCOVA — [p-value comment as in outcome 3, analysis 1]; LS Mean Difference = -0.8, 95% CI 2-sided [-3.1 to 1.5], Standard Error of Mean 1.14
Statistical Analysis 5: Comparison: Standard of Care vs Early Adalimumab; Month 18; Test type: Superiority or Other; p = 0.649, ANCOVA — [p-value comment as in outcome 3, analysis 1]; LS Mean Difference = -0.6, 95% CI 2-sided [-3.2 to 2.0], Standard Error of Mean 1.30
Statistical Analysis 6: Comparison: Standard of Care vs Early Adalimumab; Month 24; Test type: Superiority or Other; p = 0.464, ANCOVA — [p-value comment as in outcome 3, analysis 1]; LS Mean Difference = -0.8, 95% CI 2-sided [-3.0 to 1.4], Standard Error of Mean 1.11

12. Secondary Outcome: Change From Baseline in Physician's Global Assessment of Disease Activity at Months 3, 6, 9, 12, 18 and 24
Description: Physicians were asked to indicate the participant's disease activity (independent of the participant's self assessment) on a visual analogue scale (VAS) from 0 (very good) to 100 (very bad). A negative change from Baseline indicates improvement.
Time Frame: Baseline, Months 3, 6, 9, 12, 18, 24
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Standard of Care | Early Adalimumab
Number analyzed (Participants) | 35 | 38
units on a scale
  Month 3 | -29.3 (3.66) | -41.6 (3.51)
  Month 6 | -22.5 (4.25) | -48.0 (4.08)
  Month 9 | -39.6 (4.21) | -48.9 (4.04)
  Month 12 | -43.8 (4.12) | -47.3 (3.96)
  Month 18 | -45.5 (4.29) | -46.2 (4.12)
  Month 24 | -47.6 (4.23) | -47.7 (4.06)
Statistical Analysis 1: Comparison: Standard of Care vs Early Adalimumab; Month 3; Test type: Superiority or Other; p = 0.018, ANCOVA — [p-value comment as in outcome 3, analysis 1]; The a priori threshold for statistical significance is P=0.05; LS Mean Difference = -12.3, 95% CI 2-sided [-22.5 to -2.2], Standard Error of Mean 5.08
Statistical Analysis 2: Comparison: Standard of Care vs Early Adalimumab; Month 6; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; The a priori threshold for statistical significance is P=0.001; LS Mean Difference = -25.5, 95% CI 2-sided [-37.3 to -13.7], Standard Error of Mean 5.90
Statistical Analysis 3: Comparison: Standard of Care vs Early Adalimumab; Month 9; Test type: Superiority or Other; p = 0.113, ANCOVA — [p-value comment as in outcome 3, analysis 1]; LS Mean Difference = -9.4, 95% CI 2-sided [-21.0 to 2.3], Standard Error of Mean 5.84
Statistical Analysis 4: Comparison: Standard of Care vs Early Adalimumab; Month 12; Test type: Superiority or Other; p = 0.544, ANCOVA — [p-value comment as in outcome 3, analysis 1]; LS Mean Difference = -3.5, 95% CI 2-sided [-14.9 to 7.9], Standard Error of Mean 5.72
Statistical Analysis 5: Comparison: Standard of Care vs Early Adalimumab; Month 18; Test type: Superiority or Other; p = 0.916, ANCOVA — [p-value comment as in outcome 3, analysis 1]; LS Mean Difference = -0.6, 95% CI 2-sided [-12.5 to 11.2], Standard Error of Mean 5.96
Statistical Analysis 6: Comparison: Standard of Care vs Early Adalimumab; Month 24; Test type: Superiority or Other; p = 0.983, ANCOVA — [p-value comment as in outcome 3, analysis 1]; LS Mean Difference = -0.1, 95% CI 2-sided [-11.8 to 11.6], Standard Error of Mean 5.86

13. Secondary Outcome: Change From Baseline in Patient's Global Assessment of Disease Activity at Months 3, 6, 9, 12, 18 and 24
Description: Participants were asked to indicate how they were doing with their RA on a VAS from 0 (very well) to 100 (very poorly). A negative change from Baseline indicates improvement.
Time Frame: Baseline, Months 3, 6, 9, 12, 18, 24
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Standard of Care | Early Adalimumab
Number analyzed (Participants) | 35 | 38
units on a scale
  Month 3 | -19.5 (3.58) | -21.8 (3.43)
  Month 6 | -14.4 (4.05) | -19.6 (3.88)
  Month 9 | -25.4 (4.02) | -20.2 (3.86)
  Month 12 | -22.4 (3.81) | -22.3 (3.65)
  Month 18 | -29.4 (3.86) | -23.0 (3.71)
  Month 24 | -30.6 (3.99) | -23.6 (3.83)
Statistical Analysis 1: Comparison: Standard of Care vs Early Adalimumab; Month 3; Test type: Superiority or Other; p = 0.641, ANCOVA — P-values are two-sided and are based on ANCOVA model with treatment group as the fixed effect and Baseline value as the covariate; LS Mean Difference = -2.3, 95% CI 2-sided [-12.2 to 7.6], Standard Error of Mean 4.96
Statistical Analysis 2: Comparison: Standard of Care vs Early Adalimumab; Month 6; Test type: Superiority or Other; p = 0.358, ANCOVA — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = -5.2, 95% CI 2-sided [-16.4 to 6.0], Standard Error of Mean 5.61
Statistical Analysis 3: Comparison: Standard of Care vs Early Adalimumab; Month 9; Test type: Superiority or Other; p = 0.352, ANCOVA — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = 5.2, 95% CI 2-sided [-5.9 to 16.4], Standard Error of Mean 5.58
Statistical Analysis 4: Comparison: Standard of Care vs Early Adalimumab; Month 12; Test type: Superiority or Other; p = 0.990, ANCOVA — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = 0.1, 95% CI 2-sided [-10.5 to 10.6], Standard Error of Mean 5.28
Statistical Analysis 5: Comparison: Standard of Care vs Early Adalimumab; Month 18; Test type: Superiority or Other; p = 0.238, ANCOVA — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = 6.4, 95% CI 2-sided [-4.3 to 17.1], Standard Error of Mean 5.36
Statistical Analysis 6: Comparison: Standard of Care vs Early Adalimumab; Month 24; Test type: Superiority or Other; p = 0.207, ANCOVA — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = 7.1, 95% CI 2-sided [-4.0 to 18.1], Standard Error of Mean 5.54

14. Secondary Outcome: Change From Baseline in Patient's Global Assessment of Pain at Months 3, 6, 9, 12, 18 and 24
Description: Participants were asked to indicate how severe their pain had been in the previous week on a VAS from 0 (no pain) to 100 (pain as bad as it could be). A negative change from Baseline indicates improvement.
Time Frame: Baseline, Months 3, 6, 9, 12, 18, 24
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Standard of Care | Early Adalimumab
Number analyzed (Participants) | 35 | 38
units on a scale
  Month 3 | -22.0 (3.79) | -23.0 (3.64)
  Month 6 | -14.5 (3.94) | -23.0 (3.78)
  Month 9 | -21.7 (4.03) | -21.3 (3.87)
  Month 12 | -22.0 (4.01) | -24.4 (3.85)
  Month 18 | -28.1 (4.07) | -22.7 (3.90)
  Month 24 | -26.6 (4.40) | -23.6 (4.22)
Statistical Analysis 1: Comparison: Standard of Care vs Early Adalimumab; Month 3; Test type: Superiority or Other; p = 0.850, ANCOVA — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = -1.0, 95% CI 2-sided [-11.5 to 9.5], Standard Error of Mean 5.28
Statistical Analysis 2: Comparison: Standard of Care vs Early Adalimumab; Month 6; Test type: Superiority or Other; p = 0.129, ANCOVA — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = -8.4, 95% CI 2-sided [-19.4 to 2.5], Standard Error of Mean 5.49
Statistical Analysis 3: Comparison: Standard of Care vs Early Adalimumab; Month 9; Test type: Superiority or Other; p = 0.937, ANCOVA — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = 0.4, 95% CI 2-sided [-10.8 to 11.6], Standard Error of Mean 5.62
Statistical Analysis 4: Comparison: Standard of Care vs Early Adalimumab; Month 12; Test type: Superiority or Other; p = 0.670, ANCOVA — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = -2.4, 95% CI 2-sided [-13.5 to 8.8], Standard Error of Mean 5.59
Statistical Analysis 5: Comparison: Standard of Care vs Early Adalimumab; Month 18; Test type: Superiority or Other; p = 0.341, ANCOVA — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = 5.4, 95% CI 2-sided [-5.9 to 16.7], Standard Error of Mean 5.67
Statistical Analysis 6: Comparison: Standard of Care vs Early Adalimumab; Month 24; Test type: Superiority or Other; p = 0.621, ANCOVA — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = 3.0, 95% CI 2-sided [-9.2 to 15.3], Standard Error of Mean 6.13

15. Secondary Outcome: Change From Baseline in CRP at Months 3, 6, 9, 12, 18 and 24
Time Frame: Baseline, Months 3, 6, 9, 12, 18, 24
Population: Intent-to-treat population: all participants who were randomized and received at least one dose of study drug with an assessment. LOCF: missing responses were imputed by carrying forward the last non-missing post-baseline observation; n=number of participants with an assessment at given time point.
Measure: Least Squares Mean (Standard Error); unit: mg/L
Arm/Group | Standard of Care | Early Adalimumab
Number analyzed (Participants) | 35 | 38
mg/L
  Month 3; n=33, 38 | -10.2 (2.39) | -8.9 (2.23)
  Month 6; n=34, 38 | -7.6 (3.26) | -9.1 (3.08)
  Month 9; n=35, 38 | -11.3 (2.84) | -11.1 (2.72)
  Month 12; n=35, 38 | -13.7 (2.37) | -10.8 (2.28)
  Month 18; n=35, 38 | -15.2 (2.51) | -9.7 (2.41)
  Month 24; n=26, 23 | -13.5 (2.46) | -11.2 (2.36)
Statistical Analysis 1: Comparison: Standard of Care vs Early Adalimumab; Month 3; Test type: Superiority or Other; p = 0.697, ANCOVA — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = 1.3, 95% CI 2-sided [-5.3 to 7.9], Standard Error of Mean 3.29
Statistical Analysis 2: Comparison: Standard of Care vs Early Adalimumab; Month 6; Test type: Superiority or Other; p = 0.744, ANCOVA — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = -1.5, 95% CI 2-sided [-10.5 to 7.5], Standard Error of Mean 4.51
Statistical Analysis 3: Comparison: Standard of Care vs Early Adalimumab; Month 9; Test type: Superiority or Other; p = 0.967, ANCOVA — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = 0.2, 95% CI 2-sided [-7.7 to 8.0], Standard Error of Mean 3.95
Statistical Analysis 4: Comparison: Standard of Care vs Early Adalimumab; Month 12; Test type: Superiority or Other; p = 0.377, ANCOVA — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = 2.9, 95% CI 2-sided [-3.7 to 9.5], Standard Error of Mean 3.30
Statistical Analysis 5: Comparison: Standard of Care vs Early Adalimumab; Month 18; Test type: Superiority or Other; p = 0.122, ANCOVA — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = 5.5, 95% CI 2-sided [-1.5 to 12.4], Standard Error of Mean 3.50
Statistical Analysis 6: Comparison: Standard of Care vs Early Adalimumab; Month 24; Test type: Superiority or Other; p = 0.490, ANCOVA — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = 2.4, 95% CI 2-sided [-4.4 to 9.2], Standard Error of Mean 3.42

16. Secondary Outcome: Change From Baseline in Disease Activity Score DAS28(CRP) at Months 3, 6, 9, 12, 18 and 24
Description: The DAS28 is a validated index of rheumatoid arthritis disease activity. Twenty-eight tender joint counts, 28 swollen joint counts, CRP, and general health are included in the DAS28 score. Scores on the DAS28 range from 0 to 10, with higher scores indicating higher disease activity.
Time Frame: Baseline, Months 3, 6, 9, 12, 18, 24
Population: as for outcome 15
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Standard of Care | Early Adalimumab
Number analyzed (Participants) | 35 | 38
units on a scale
  Month 3; n=33, 38 | -1.4 (0.20) | -1.8 (0.18)
  Month 6; n=34, 38 | -1.4 (0.21) | -2.3 (0.20)
  Month 9; n=35, 38 | -2.0 (0.21) | -2.3 (0.20)
  Month 12; n=35, 38 | -2.1 (0.20) | -2.4 (0.19)
  Month 18; n=35, 38 | -2.4 (0.22) | -2.4 (0.21)
  Month 24; n=35, 38 | -2.6 (0.20) | -2.6 (0.19)
Statistical Analysis 1: Comparison: Standard of Care vs Early Adalimumab; Month 3; Test type: Superiority or Other; p = 0.102, ANCOVA — [p-value comment as in outcome 3, analysis 1]; LS Mean Difference = -0.4, 95% CI 2-sided [-1.0 to 0.1], Standard Error of Mean 0.27
Statistical Analysis 2: Comparison: Standard of Care vs Early Adalimumab; Month 6; Test type: Superiority or Other; p = 0.003, ANCOVA — [p-value comment as in outcome 3, analysis 1]; The a priori threshold for statistical significance is P=0.01; LS Mean Difference = -0.9, 95% CI 2-sided [-1.5 to -0.3], Standard Error of Mean 0.29
Statistical Analysis 3: Comparison: Standard of Care vs Early Adalimumab; Month 9; Test type: Superiority or Other; p = 0.214, ANCOVA — [p-value comment as in outcome 3, analysis 1]; LS Mean Difference = -0.4, 95% CI 2-sided [-0.9 to 0.2], Standard Error of Mean 0.29
Statistical Analysis 4: Comparison: Standard of Care vs Early Adalimumab; Month 12; Test type: Superiority or Other; p = 0.339, ANCOVA — [p-value comment as in outcome 3, analysis 1]; LS Mean Difference = -0.3, 95% CI 2-sided [-0.8 to 0.3], Standard Error of Mean 0.27
Statistical Analysis 5: Comparison: Standard of Care vs Early Adalimumab; Month 18; Test type: Superiority or Other; p = 0.973, ANCOVA — [p-value comment as in outcome 3, analysis 1]; LS Mean Difference = 0.0, 95% CI 2-sided [-0.6 to 0.6], Standard Error of Mean 0.30
Statistical Analysis 6: Comparison: Standard of Care vs Early Adalimumab; Month 24; Test type: Superiority or Other; p = 0.755, ANCOVA — [p-value comment as in outcome 3, analysis 1]; LS Mean Difference = -0.1, 95% CI 2-sided [-0.6 to 0.5], Standard Error of Mean 0.28

17. Secondary Outcome: Percentage of Participants With DAS28(CRP) Remission at Months 3, 6, 9, 12, 18 and 24
Description: DAS28(CRP) remission was defined as DAS28(CRP) < 2.6. The DAS28(CRP) is a validated index of rheumatoid arthritis disease activity. Twenty-eight tender joint counts, 28 swollen joint counts, CRP, and general health are included in the DAS28 score. Scores on the DAS28 range from 0 to 10, with higher scores indicating higher disease activity.
Time Frame: Months 3, 6, 9, 12, 18, 24
Population: Intent-to-treat population: all participants who were randomized and received at least one dose of study drug with an assessment (non-responder imputation).
Measure: Number; unit: percentage of participants
Arm/Group | Standard of Care | Early Adalimumab
Number analyzed (Participants) | 35 | 39
percentage of participants
  Month 3 | 8.6 | 17.9
  Month 6 | 11.4 | 35.9
  Month 9 | 31.4 | 28.2
  Month 12 | 22.9 | 35.9
  Month 18 | 34.3 | 30.8
  Month 24 | 42.9 | 38.5
Statistical Analysis 1: Comparison: Standard of Care vs Early Adalimumab; Month 3; Test type: Superiority or Other; p = 0.316, Fisher Exact; Two-sided Fisher Exact test; Difference in percentage = 9.4, 95% CI 2-sided [-7.09 to 25.13]
Statistical Analysis 2: Comparison: Standard of Care vs Early Adalimumab; Month 6; Test type: Superiority or Other; p = 0.014, Chi-squared; P-value is based on two-sided Pearson's chi-square test. The a priori threshold for statistical significance is P=0.05; Difference in percentage = 24.5, 95% CI 2-sided [6.09 to 42.85]
Statistical Analysis 3: Comparison: Standard of Care vs Early Adalimumab; Month 9; Test type: Superiority or Other; p = 0.762, Chi-squared; P-value is based on two-sided Pearson's chi-square test; Difference in percentage = -3.2, 95% CI 2-sided [-24.10 to 17.66]
Statistical Analysis 4: Comparison: Standard of Care vs Early Adalimumab; Month 12; Test type: Superiority or Other; p = 0.220, Chi-squared; P-value is based on two-sided Pearson's chi-square test; Difference in percentage = 13.0, 95% CI 2-sided [-7.46 to 33.54]
Statistical Analysis 5: Comparison: Standard of Care vs Early Adalimumab; Month 18; Test type: Superiority or Other; p = 0.747, Chi-squared; P-value is based on two-sided Pearson's chi-square test; Difference in percentage = -3.5, 95% CI 2-sided [-24.90 to 17.86]
Statistical Analysis 6: Comparison: Standard of Care vs Early Adalimumab; Month 24; Test type: Superiority or Other; p = 0.701, Chi-squared; P-value is based on two-sided Pearson's chi-square test; Difference in percentage = -4.4, 95% CI 2-sided [-26.80 to 18.01]

18. Secondary Outcome: Percentage of Participants With DAS28(CRP) Low Disease Activity at Months 3, 6, 9, 12, 18 and 24
Description: DAS28(CRP) low disease activity was defined as DAS28(CRP) < 3.2. The DAS28(CRP) is a validated index of rheumatoid arthritis disease activity. Twenty-eight tender joint counts, 28 swollen joint counts, CRP, and general health are included in the DAS28 score. Scores on the DAS28 range from 0 to 10, with higher scores indicating higher disease activity.
Time Frame: Months 3, 6, 9, 12, 18, 24
Population: as for outcome 17
Measure: Number; unit: percentage of participants
Arm/Group | Standard of Care | Early Adalimumab
Number analyzed (Participants) | 35 | 39
percentage of participants
  Month 3 | 22.9 | 33.3
  Month 6 | 28.6 | 51.3
  Month 9 | 51.4 | 56.4
  Month 12 | 48.6 | 56.4
  Month 18 | 51.4 | 48.7
  Month 24 | 54.3 | 43.6
Statistical Analysis 1: Comparison: Standard of Care vs Early Adalimumab; Month 3; Test type: Superiority or Other; p = 0.318, Chi-squared; P-value is based on two-sided Pearson's chi-square test; Difference in percentage = 10.5, 95% CI 2-sided [-9.83 to 30.78]
Statistical Analysis 2: Comparison: Standard of Care vs Early Adalimumab; Month 6; Test type: Superiority or Other; p = 0.047, Chi-squared; P-value is based on two-sided Pearson's chi-square test. The a priori threshold for statistical significance is P=0.05; Difference in percentage = 22.7, 95% CI 2-sided [1.03 to 44.39]
Statistical Analysis 3: Comparison: Standard of Care vs Early Adalimumab; Month 9; Test type: Superiority or Other; p = 0.668, Chi-squared; P-value is based on two-sided Pearson's chi-square test; Difference in percentage = 5.0, 95% CI 2-sided [-17.74 to 27.71]
Statistical Analysis 4: Comparison: Standard of Care vs Early Adalimumab; Month 12; Test type: Superiority or Other; p = 0.500, Chi-squared; P-value is based on two-sided Pearson's chi-square test; Difference in percentage = 7.8, 95% CI 2-sided [-14.88 to 30.56]
Statistical Analysis 5: Comparison: Standard of Care vs Early Adalimumab; Month 18; Test type: Superiority or Other; p = 0.816, Chi-squared; P-value is based on two-sided Pearson's chi-square test; Difference in percentage = -2.7, 95% CI 2-sided [-25.52 to 20.10]
Statistical Analysis 6: Comparison: Standard of Care vs Early Adalimumab; Month 24; Test type: Superiority or Other; p = 0.358, Chi-squared; P-value is based on two-sided Pearson's chi-square test; Difference in percentage = -10.7, 95% CI 2-sided [-33.38 to 11.99]

19. Secondary Outcome: Percentage of Participants With European League Against Rheumatism (EULAR) Good Response at Months 3, 6, 9, 12, 18 and 24
Description: A EULAR response reflects an improvement in disease activity and an attainment of a lower degree of disease activity based on the DAS28 score. The DAS28 score ranges from 0-10, with higher scores indicating more disease activity. A Good EULAR Response is defined as an improvement (decrease) in the DAS28 of ≥ 1.2 compared with Baseline and attainment of a DAS28 score of ≤ 3.2.
Time Frame: Months 3, 6, 9, 12, 18, 24
Population: as for outcome 17
Measure: Number; unit: percentage of participants
Arm/Group | Standard of Care | Early Adalimumab
Number analyzed (Participants) | 35 | 39
percentage of participants
  Month 3 | 22.9 | 30.8
  Month 6 | 28.6 | 48.7
  Month 9 | 48.6 | 51.3
  Month 12 | 45.7 | 53.8
  Month 18 | 51.4 | 48.7
  Month 24 | 54.3 | 43.6
Statistical Analysis 1: Comparison: Standard of Care vs Early Adalimumab; Month 3; Test type: Superiority or Other; p = 0.444, Chi-squared; P-value is based on two-sided Pearson's chi-square test; Difference in percentage = 7.9, 95% CI 2-sided [-12.17 to 28.00]
Statistical Analysis 2: Comparison: Standard of Care vs Early Adalimumab; Month 6; Test type: Superiority or Other; p = 0.076, Chi-squared; P-value is based on two-sided Pearson's chi-square test; Difference in percentage = 20.1, 95% CI 2-sided [-1.53 to 41.83]
Statistical Analysis 3: Comparison: Standard of Care vs Early Adalimumab; Month 9; Test type: Superiority or Other; p = 0.816, Chi-squared; P-value is based on two-sided Pearson's chi-square test; Difference in percentage = 2.7, 95% CI 2-sided [-20.10 to 25.52]
Statistical Analysis 4: Comparison: Standard of Care vs Early Adalimumab; Month 12; Test type: Superiority or Other; p = 0.485, Chi-squared; P-value is based on two-sided Pearson's chi-square test; Difference in percentage = 8.1, 95% CI 2-sided [-14.61 to 30.87]
Statistical Analysis 5: Comparison: Standard of Care vs Early Adalimumab; Month 18; Test type: Superiority or Other; p = 0.816, Chi-squared; P-value is based on two-sided Pearson's chi-square test; Difference in percentage = -2.7, 95% CI 2-sided [-25.52 to 20.10]
Statistical Analysis 6: Comparison: Standard of Care vs Early Adalimumab; Month 24; Test type: Superiority or Other; p = 0.358, Chi-squared; P-value is based on two-sided Pearson's chi-square test; Difference in percentage = -10.7, 95% CI 2-sided [-33.38 to 11.99]

20. Secondary Outcome: Percentage of Participants With EULAR Moderate Response at Months 3, 6, 9, 12, 18 and 24
Description: A EULAR response reflects an improvement in disease activity and an attainment of a lower degree of disease activity based on the DAS28 score. The DAS28 score ranges from 0-10, with higher scores indicating more disease activity. A Moderate EULAR Response is defined as either: an improvement (decrease) in the DAS28 of > 0.6 and < 1.2 from Baseline and attainment of a DAS28 score of ≤ 5.1; or an improvement (decrease) in the DAS28 of ≥ 1.2 from Baseline and attainment of a DAS28 score of > 3.2.
Time Frame: Months 3, 6, 9, 12, 18, 24
Population: as for outcome 17
Measure: Number; unit: percentage of participants
Arm/Group | Standard of Care | Early Adalimumab
Number analyzed (Participants) | 35 | 39
percentage of participants
  Month 3 | 37.1 | 48.7
  Month 6 | 25.7 | 30.8
  Month 9 | 28.6 | 28.2
  Month 12 | 37.1 | 23.1
  Month 18 | 22.9 | 10.3
  Month 24 | 14.3 | 10.3
Statistical Analysis 1: Comparison: Standard of Care vs Early Adalimumab; Month 3; Test type: Superiority or Other; p = 0.316, Chi-squared; P-value is based on two-sided Pearson's chi-square test; Difference in percentage = 11.6, 95% CI 2-sided [-10.84 to 33.99]
Statistical Analysis 2: Comparison: Standard of Care vs Early Adalimumab; Month 6; Test type: Superiority or Other; p = 0.630, Chi-squared; P-value is based on two-sided Pearson's chi-square test; Difference in percentage = 5.1, 95% CI 2-sided [-15.43 to 25.54]
Statistical Analysis 3: Comparison: Standard of Care vs Early Adalimumab; Month 9; Test type: Superiority or Other; p = 0.972, Chi-squared; P-value is based on two-sided Pearson's chi-square test; Difference in percentage = -0.4, 95% CI 2-sided [-20.94 to 20.21]
Statistical Analysis 4: Comparison: Standard of Care vs Early Adalimumab; Month 12; Test type: Superiority or Other; p = 0.186, Chi-squared; P-value is based on two-sided Pearson's chi-square test; Difference in percentage = -14.1, 95% CI 2-sided [-34.83 to 6.70]
Statistical Analysis 5: Comparison: Standard of Care vs Early Adalimumab; Month 18; Test type: Superiority or Other; p = 0.142, Chi-squared; P-value is based on two-sided Pearson's chi-square test; Difference in percentage = -12.6, 95% CI 2-sided [-29.46 to 4.26]
Statistical Analysis 6: Comparison: Standard of Care vs Early Adalimumab; Month 24; Test type: Superiority or Other; p = 0.727, Chi-squared; P-value is based on two-sided Pearson's chi-square test; Difference in percentage = -4.0, 95% CI 2-sided [-20.34 to 11.52]

21. Secondary Outcome: Percentage of Participants With Flare-Up After Remission by Month 24
Description: Percentage of participants with a flare-up after remission by Month 24, defined as participants who reached remission (DAS28 < 2.6) but later had two consecutive visits with DAS28 ≥ 2.6 (based on observed cases only). The DAS28 is a validated index of rheumatoid arthritis disease activity. Twenty-eight tender joint counts, 28 swollen joint counts, CRP, and general health are included in the DAS28 score. Scores on the DAS28 range from 0 to 10, with higher scores indicating higher disease activity.
Time Frame: Month 24
Population: Intent-to-treat population: all participants who were randomized and received at least one dose of study drug and had an assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Standard of Care | Early Adalimumab
Number analyzed (Participants) | 35 | 39
percentage of participants | 8.6 | 15.4
Statistical Analysis 1: Comparison: Standard of Care vs Early Adalimumab; Test type: Superiority or Other; p = 0.486, Fisher Exact; Two-sided Fisher Exact test; Difference in percentage = 6.8, 95% CI 2-sided [-9.21 to 22.22]

22. Secondary Outcome: Change From Baseline in Disability Index of the Health Assessment Questionnaire (HAQ-DI) at Months 3, 6, 9, 12, 18 and 24
Description: HAQ is a participant-reported questionnaire specific for rheumatoid arthritis. It consists of 20 questions referring to eight domains: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and daily activities. Participants assessed their ability to do each task over the past week using the following response categories: without any difficulty (0); with some difficulty (1); with much difficulty (2); and unable to do (3). Scores on each task were summed and averaged to provide an overall score ranging from 0 to 3, where zero represents no disability and three very severe, high-dependency disability. A lower HAQ-DI score is better.
Time Frame: Baseline, Months 3, 6, 9, 12, 18, 24
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Standard of Care | Early Adalimumab
Number analyzed (Participants) | 35 | 38
units on a scale
  Month 3 | -0.41 (0.094) | -0.38 (0.090)
  Month 6 | -0.29 (0.095) | -0.46 (0.092)
  Month 9 | -0.52 (0.095) | -0.50 (0.092)
  Month 12 | -0.60 (0.093) | -0.50 (0.089)
  Month 18 | -0.60 (0.102) | -0.55 (0.098)
  Month 24 | -0.61 (0.107) | -0.53 (0.102)
Statistical Analysis 1: Comparison: Standard of Care vs Early Adalimumab; Month 3; Test type: Superiority or Other; p = 0.809, ANCOVA — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = 0.03, 95% CI 2-sided [-0.23 to 0.29], Standard Error of Mean 0.130
Statistical Analysis 2: Comparison: Standard of Care vs Early Adalimumab; Month 6; Test type: Superiority or Other; p = 0.194, ANCOVA — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = -0.17, 95% CI 2-sided [-0.44 to 0.09], Standard Error of Mean 0.132
Statistical Analysis 3: Comparison: Standard of Care vs Early Adalimumab; Month 9; Test type: Superiority or Other; p = 0.863, ANCOVA — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = 0.02, 95% CI 2-sided [-0.24 to 0.29], Standard Error of Mean 0.132
Statistical Analysis 4: Comparison: Standard of Care vs Early Adalimumab; Month 12; Test type: Superiority or Other; p = 0.452, ANCOVA — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = 0.10, 95% CI 2-sided [-0.16 to 0.35], Standard Error of Mean 0.129
Statistical Analysis 5: Comparison: Standard of Care vs Early Adalimumab; Month 18; Test type: Superiority or Other; p = 0.738, ANCOVA — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = 0.05, 95% CI 2-sided [-0.23 to 0.33], Standard Error of Mean 0.141
Statistical Analysis 6: Comparison: Standard of Care vs Early Adalimumab; Month 24; Test type: Superiority or Other; p = 0.572, ANCOVA — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = 0.08, 95% CI 2-sided [-0.21 to 0.38], Standard Error of Mean 0.148

23. Secondary Outcome: Percentage of Participants Achieving Minimal Clinical Important Difference (MCID) in HAQ at Months 3, 6, 9, 12, 18 and 24
Description: The percentage of participants achieving MCID in HAQ, defined as a 0.22 unit decrease in HAQ. HAQ is a participant-reported questionnaire specific for rheumatoid arthritis. It consists of 20 questions referring to eight domains: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and daily activities. Participants assessed their ability to do each task over the past week using the following response categories: without any difficulty (0); with some difficulty (1); with much difficulty (2); and unable to do (3). Scores on each task were summed and averaged to provide an overall score ranging from 0 to 3, where zero represents no disability and three very severe, high-dependency disability. A lower HAQ-DI score is better.
Time Frame: Months 3, 6, 9, 12, 18, 24
Population: as for outcome 17
Measure: Number; unit: percentage of participants
Arm/Group | Standard of Care | Early Adalimumab
Number analyzed (Participants) | 35 | 39
percentage of participants
  Month 3 | 65.7 | 53.8
  Month 6 | 54.3 | 51.3
  Month 9 | 57.1 | 64.1
  Month 12 | 68.6 | 59.0
  Month 18 | 57.1 | 53.8
  Month 24 | 57.1 | 41.0
Statistical Analysis 1: Comparison: Standard of Care vs Early Adalimumab; Month 3; Test type: Superiority or Other; p = 0.299, Chi-squared; P-value is based on two-sided Pearson's chi-square test; Difference in percentage = -11.9, 95% CI 2-sided [-34.05 to 10.31]
Statistical Analysis 2: Comparison: Standard of Care vs Early Adalimumab; Month 6; Test type: Superiority or Other; p = 0.796, Chi-squared; P-value is based on two-sided Pearson's chi-square test; Difference in percentage = -3.0, 95% CI 2-sided [-25.77 to 19.77]
Statistical Analysis 3: Comparison: Standard of Care vs Early Adalimumab; Month 9; Test type: Superiority or Other; p = 0.540, Chi-squared; P-value is based on two-sided Pearson's chi-square test; Difference in percentage = 7.0, 95% CI 2-sided [-15.30 to 29.22]
Statistical Analysis 4: Comparison: Standard of Care vs Early Adalimumab; Month 12; Test type: Superiority or Other; p = 0.392, Chi-squared; P-value is based on two-sided Pearson's chi-square test; Difference in percentage = -9.6, 95% CI 2-sided [-31.39 to 12.19]
Statistical Analysis 5: Comparison: Standard of Care vs Early Adalimumab; Month 18; Test type: Superiority or Other; p = 0.776, Chi-squared; P-value is based on two-sided Pearson's chi-square test; Difference in percentage = -3.3, 95% CI 2-sided [-25.96 to 19.37]
Statistical Analysis 6: Comparison: Standard of Care vs Early Adalimumab; Month 24; Test type: Superiority or Other; p = 0.166, Chi-squared; P-value is based on two-sided Pearson's chi-square test; Difference in percentage = -16.1, 95% CI 2-sided [-38.64 to 6.40]

24. Secondary Outcome: Percentage of Participants Achieving HAQ < 0.5 at Months 3, 6, 9, 12, 18 and 24
Description: The percentage of participants achieving HAQ < 0.5. HAQ is a participant-reported questionnaire specific for rheumatoid arthritis. It consists of 20 questions referring to eight domains: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and daily activities. Participants assessed their ability to do each task over the past week using the following response categories: without any difficulty (0); with some difficulty (1); with much difficulty (2); and unable to do (3). Scores on each task were summed and averaged to provide an overall score ranging from 0 to 3, where zero represents no disability and three very severe, high-dependency disability. HAQ remission indicating normal physical function is defined by HAQ-DI < 0.5. A lower HAQ-DI score is better.
Time Frame: Months 3, 6, 9, 12, 18, 24
Population: as for outcome 17
Measure: Number; unit: percentage of participants
Arm/Group | Standard of Care | Early Adalimumab
Number analyzed (Participants) | 35 | 39
percentage of participants
  Month 3 | 31.4 | 20.5
  Month 6 | 22.9 | 30.8
  Month 9 | 34.3 | 35.9
  Month 12 | 34.3 | 33.3
  Month 18 | 28.6 | 30.8
  Month 24 | 28.6 | 30.8
Statistical Analysis 1: Comparison: Standard of Care vs Early Adalimumab; Month 3; Test type: Superiority or Other; p = 0.283, Chi-squared; P-value is based on two-sided Pearson's chi-square test; Difference in percentage = -10.9, 95% CI 2-sided [-30.84 to 9.01]
Statistical Analysis 2: Comparison: Standard of Care vs Early Adalimumab; Month 6; Test type: Superiority or Other; p = 0.444, Chi-squared; P-value is based on two-sided Pearson's chi-square test; Difference in percentage = 7.9, 95% CI 2-sided [-12.17 to 28.00]
Statistical Analysis 3: Comparison: Standard of Care vs Early Adalimumab; Month 9; Test type: Superiority or Other; p = 0.885, Chi-squared; P-value is based on two-sided Pearson's chi-square test; Difference in percentage = 1.6, 95% CI 2-sided [-20.16 to 23.38]
Statistical Analysis 4: Comparison: Standard of Care vs Early Adalimumab; Month 12; Test type: Superiority or Other; p = 0.931, Chi-squared; P-value is based on two-sided Pearson's chi-square test; Difference in percentage = -1.0, 95% CI 2-sided [-22.54 to 20.64]
Statistical Analysis 5: Comparison: Standard of Care vs Early Adalimumab; Month 18; Test type: Superiority or Other; p = 0.836, Chi-squared; P-value is based on two-sided Pearson's chi-square test; Difference in percentage = 2.2, 95% CI 2-sided [-18.63 to 23.03]
Statistical Analysis 6: Comparison: Standard of Care vs Early Adalimumab; Month 24; Test type: Superiority or Other; p = 0.836, Chi-squared; P-value is based on two-sided Pearson's chi-square test; Difference in percentage = 2.2, 95% CI 2-sided [-18.63 to 23.03]

25. Secondary Outcome: Change From Baseline in Functional Assessment of Chronic Illness Therapy (FACIT) Fatigue Scale at Months 3, 6, 9, 12, 18 and 24
Description: The FACIT-Fatigue questionnaire is a self-administered patient questionnaire that consists of 13 questions designed to measure the degree of fatigue experienced by participants in the previous 7 days. Participants respond to the questions on a scale from 'not at all' (0) to 'very much' (4). The scale score is computed by summing the item scores, after reversing those items that are worded in the negative direction. The FACIT-Fatigue subscale score ranges from 0 to 52, where higher scores represent less fatigue.
Time Frame: Baseline, Months 3, 6, 9, 12, 18, 24
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Standard of Care | Early Adalimumab
Number analyzed (Participants) | 35 | 38
units on a scale
  Month 3 | 7.1 (1.62) | 8.0 (1.56)
  Month 6 | 5.4 (1.77) | 8.2 (1.70)
  Month 9 | 9.5 (1.70) | 8.0 (1.63)
  Month 12 | 10.7 (1.80) | 8.0 (1.73)
  Month 18 | 10.2 (1.98) | 8.2 (1.90)
  Month 24 | 9.8 (2.00) | 8.8 (1.92)
Statistical Analysis 1: Comparison: Standard of Care vs Early Adalimumab; Month 3; Test type: Superiority or Other; p = 0.699, ANCOVA — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = 0.9, 95% CI 2-sided [-3.6 to 5.4], Standard Error of Mean 2.25
Statistical Analysis 2: Comparison: Standard of Care vs Early Adalimumab; Month 6; Test type: Superiority or Other; p = 0.261, ANCOVA — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = 2.8, 95% CI 2-sided [-2.1 to 7.7], Standard Error of Mean 2.45
Statistical Analysis 3: Comparison: Standard of Care vs Early Adalimumab; Month 9; Test type: Superiority or Other; p = 0.514, ANCOVA — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = -1.5, 95% CI 2-sided [-6.2 to 3.2], Standard Error of Mean 2.36
Statistical Analysis 4: Comparison: Standard of Care vs Early Adalimumab; Month 12; Test type: Superiority or Other; p = 0.283, ANCOVA — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = -2.7, 95% CI 2-sided [-7.7 to 2.3], Standard Error of Mean 2.50
Statistical Analysis 5: Comparison: Standard of Care vs Early Adalimumab; Month 18; Test type: Superiority or Other; p = 0.461, ANCOVA — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = -2.0, 95% CI 2-sided [-7.5 to 3.4], Standard Error of Mean 2.75
Statistical Analysis 6: Comparison: Standard of Care vs Early Adalimumab; Month 24; Test type: Superiority or Other; p = 0.703, ANCOVA — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = -1.1, 95% CI 2-sided [-6.6 to 4.5], Standard Error of Mean 2.78

26. Secondary Outcome: Percentage of Participants Achieving MCID in FACIT-Fatigue Scale at Months 3, 6, 9, 12, 18 and 24
Description: The FACIT-Fatigue questionnaire is a self-administered patient questionnaire that consists of 13 questions designed to measure the degree of fatigue experienced by participants in the previous 7 days. Participants respond to the questions on a scale from 'not at all' (0) to 'very much' (4). The scale score is computed by summing the item scores, after reversing those items that are worded in the negative direction. The FACIT-Fatigue subscale score ranges from 0 to 52, where higher scores represent less fatigue. The MCID was defined as a 3.56-unit decrease in FACIT-Fatigue Scale.
Time Frame: Months 3, 6, 9, 12, 18, 24
Population: as for outcome 17
Measure: Number; unit: percentage of participants
Arm/Group | Standard of Care | Early Adalimumab
Number analyzed (Participants) | 35 | 38
percentage of participants
  Month 3 | 14.3 | 13.2
  Month 6 | 14.3 | 7.9
  Month 9 | 17.1 | 5.3
  Month 12 | 8.6 | 13.2
  Month 18 | 8.6 | 15.8
  Month 24 | 11.4 | 5.3
Statistical Analysis 1: Comparison: Standard of Care vs Early Adalimumab; Month 3; Test type: Superiority or Other; p = 1.000, Fisher Exact; Two-sided Fisher Exact test; Difference in percentage = -1.1, 95% CI 2-sided [-17.94 to 15.16]
Statistical Analysis 2: Comparison: Standard of Care vs Early Adalimumab; Month 6; Test type: Superiority or Other; p = 0.468, Fisher Exact; Two-sided Fisher Exact test; Difference in percentage = -6.4, 95% CI 2-sided [-22.34 to 8.81]
Statistical Analysis 3: Comparison: Standard of Care vs Early Adalimumab; Month 9; Test type: Superiority or Other; p = 0.142, Fisher Exact; Two-sided Fisher Exact test; Difference in percentage = -11.9, 95% CI 2-sided [-27.88 to 3.16]
Statistical Analysis 4: Comparison: Standard of Care vs Early Adalimumab; Month 12; Test type: Superiority or Other; p = 0.712, Fisher Exact; Two-sided Fisher Exact test; Difference in percentage = 4.6, 95% CI 2-sided [-11.08 to 19.83]
Statistical Analysis 5: Comparison: Standard of Care vs Early Adalimumab; Month 18; Test type: Superiority or Other; p = 0.482, Fisher Exact; Two-sided Fisher Exact test; Difference in percentage = 7.2, 95% CI 2-sided [-8.92 to 22.89]
Statistical Analysis 6: Comparison: Standard of Care vs Early Adalimumab; Month 24; Test type: Superiority or Other; p = 0.418, Fisher Exact; Two-sided Fisher Exact test; Difference in percentage = -6.2, 95% CI 2-sided [-21.18 to 7.69]

27. Secondary Outcome: Change From Baseline in Work Limitations Questionnaire (WLQ) at Months 3, 6, 9, 12, 18 and 24
Description: The WLQ was used to measure the impairment in work-related productivity, with reference to the previous two weeks. Each work-related question is scored from 0 to 4 and the total score ranges from 0-100, with lower scores signifying fewer limitations at work.
Time Frame: Baseline, Months 3, 6, 9, 12, 18, 24
Population: Intent-to-treat population: all participants who were randomized and received at least one dose of study drug. LOCF: missing responses were imputed by carrying forward the last non-missing post-baseline observation; n=number of participants with an assessment at given time point.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Standard of Care | Early Adalimumab
Number analyzed (Participants) | 35 | 39
units on a scale
  Month 3; n=23, 24 | -7.0 (4.18) | -11.5 (4.10)
  Month 6; n=24, 25 | -6.1 (4.20) | -13.9 (4.11)
  Month 9; n=25, 25 | -8.4 (4.45) | -11.8 (4.45)
  Month 12; n=25, 25 | -15.2 (4.05) | -11.8 (4.05)
  Month 18; n=25, 25 | -15.6 (4.51) | -12.8 (4.51)
  Month 24; n=25, 25 | -13.7 (4.34) | -12.6 (4.34)
Statistical Analysis 1: Comparison: Standard of Care vs Early Adalimumab; Month 3; Test type: Superiority or Other; p = 0.453, ANCOVA — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = -4.4, 95% CI 2-sided [-16.3 to 7.4], Standard Error of Mean 5.86
Statistical Analysis 2: Comparison: Standard of Care vs Early Adalimumab; Month 6; Test type: Superiority or Other; p = 0.187, ANCOVA — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = -7.9, 95% CI 2-sided [-19.7 to 4.0], Standard Error of Mean 5.88
Statistical Analysis 3: Comparison: Standard of Care vs Early Adalimumab; Month 9; Test type: Superiority or Other; p = 0.598, ANCOVA — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = -3.4, 95% CI 2-sided [-16.1 to 9.4], Standard Error of Mean 6.31
Statistical Analysis 4: Comparison: Standard of Care vs Early Adalimumab; Month 12; Test type: Superiority or Other; p = 0.558, ANCOVA — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = 3.4, 95% CI 2-sided [-8.2 to 15.0], Standard Error of Mean 5.75
Statistical Analysis 5: Comparison: Standard of Care vs Early Adalimumab; Month 18; Test type: Superiority or Other; p = 0.669, ANCOVA — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = 2.7, 95% CI 2-sided [-10.1 to 15.6], Standard Error of Mean 6.40
Statistical Analysis 6: Comparison: Standard of Care vs Early Adalimumab; Month 24; Test type: Superiority or Other; p = 0.865, ANCOVA — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = 1.1, 95% CI 2-sided [-11.3 to 13.5], Standard Error of Mean 6.16

28. Secondary Outcome: Change From Baseline in EuroQOL Questionnaire (EQ-5D) Index Score at Months 3, 6, 9, 12, 18 and 24
Description: The EQ-5D is a participant answered questionnaire scoring 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. EQ-5D health states, defined by the EQ-5D descriptive system, are converted into a single summary index by applying a formula that essentially attaches values (also called QOL weights or QOL utilities) to each of the levels in each dimension. EQ-5D Summary Index values range from -0.594 to 1 (with higher scores indicating better health state).
Time Frame: Baseline, Months 3, 6, 9, 12, 18, 24
Population: as for outcome 27
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Standard of Care | Early Adalimumab
Number analyzed (Participants) | 35 | 39
units on a scale
  Month 3; n=34, 34 | 0.21 (0.041) | 0.22 (0.041)
  Month 6; n=35, 36 | 0.18 (0.044) | 0.23 (0.044)
  Month 9; n=35, 36 | 0.26 (0.044) | 0.22 (0.044)
  Month 12; n=35, 36 | 0.25 (0.040) | 0.26 (0.040)
  Month 18; n=35, 36 | 0.25 (0.045) | 0.24 (0.045)
  Month 24; n=35, 36 | 0.26 (0.049) | 0.22 (0.049)
Statistical Analysis 1: Comparison: Standard of Care vs Early Adalimumab; Month 3; Test type: Superiority or Other; p = 0.809, ANCOVA — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = 0.01, 95% CI 2-sided [-0.10 to 0.13], Standard Error of Mean 0.058
Statistical Analysis 2: Comparison: Standard of Care vs Early Adalimumab; Month 6; Test type: Superiority or Other; p = 0.447, ANCOVA — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = 0.05, 95% CI 2-sided [-0.08 to 0.17], Standard Error of Mean 0.062
Statistical Analysis 3: Comparison: Standard of Care vs Early Adalimumab; Month 9; Test type: Superiority or Other; p = 0.579, ANCOVA — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = -0.03, 95% CI 2-sided [-0.16 to 0.09], Standard Error of Mean 0.062
Statistical Analysis 4: Comparison: Standard of Care vs Early Adalimumab; Month 12; Test type: Superiority or Other; p = 0.922, ANCOVA — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = 0.01, 95% CI 2-sided [-0.11 to 0.12], Standard Error of Mean 0.057
Statistical Analysis 5: Comparison: Standard of Care vs Early Adalimumab; Month 18; Test type: Superiority or Other; p = 0.894, ANCOVA — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = -0.01, 95% CI 2-sided [-0.14 to 0.12], Standard Error of Mean 0.064
Statistical Analysis 6: Comparison: Standard of Care vs Early Adalimumab; Month 24; Test type: Superiority or Other; p = 0.611, ANCOVA — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = -0.04, 95% CI 2-sided [-0.17 to 0.10], Standard Error of Mean 0.070

29. Secondary Outcome: Change From Baseline in EQ-5D VAS at Months 3, 6, 9, 12, 18 and 24
Description: The EQ-5D VAS records the participant's self-rated health on a scale from 0-100 where 100 is the 'best imaginable health state' and 0 is the 'worst imaginable health state.'
Time Frame: Baseline, Months 3, 6, 9, 12, 18, 24
Population: Intent-to-treat population: all participants who were randomized and received at least one dose of study drug and had an assessment. LOCF: missing responses were imputed by carrying forward the last non-missing post-baseline observation.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Standard of Care | Early Adalimumab
Number analyzed (Participants) | 35 | 38
units on a scale
  Month 3 | 18.7 (3.18) | 16.2 (3.05)
  Month 6 | 10.7 (3.70) | 18.6 (3.55)
  Month 9 | 20.1 (3.78) | 17.7 (3.63)
  Month 12 | 22.2 (3.46) | 19.5 (3.32)
  Month 18 | 22.3 (3.62) | 21.2 (3.47)
  Month 24 | 22.1 (4.11) | 19.7 (3.95)
Statistical Analysis 1: Comparison: Standard of Care vs Early Adalimumab; Month 3; Test type: Superiority or Other; p = 0.572, ANCOVA — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = -2.5, 95% CI 2-sided [-11.3 to 6.3], Standard Error of Mean 4.42
Statistical Analysis 2: Comparison: Standard of Care vs Early Adalimumab; Month 6; Test type: Superiority or Other; p = 0.130, ANCOVA — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = 7.9, 95% CI 2-sided [-2.4 to 18.2], Standard Error of Mean 5.15
Statistical Analysis 3: Comparison: Standard of Care vs Early Adalimumab; Month 9; Test type: Superiority or Other; p = 0.649, ANCOVA — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = -2.4, 95% CI 2-sided [-12.9 to 8.1], Standard Error of Mean 5.26
Statistical Analysis 4: Comparison: Standard of Care vs Early Adalimumab; Month 12; Test type: Superiority or Other; p = 0.579, ANCOVA — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = -2.7, 95% CI 2-sided [-12.3 to 6.9], Standard Error of Mean 4.80
Statistical Analysis 5: Comparison: Standard of Care vs Early Adalimumab; Month 18; Test type: Superiority or Other; p = 0.826, ANCOVA — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = -1.1, 95% CI 2-sided [-11.1 to 8.9], Standard Error of Mean 5.03
Statistical Analysis 6: Comparison: Standard of Care vs Early Adalimumab; Month 24; Test type: Superiority or Other; p = 0.675, ANCOVA — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = -2.4, 95% CI 2-sided [-13.8 to 9.0], Standard Error of Mean 5.72

30. Secondary Outcome: Change From Baseline in Beck Depression Inventory (BDI-II) Scores at Months 3, 6, 9, 12, 18 and 24
Description: BDI is a 21-item questionnaire, participant self-report rating inventory that measures characteristic attitudes and symptoms of depression. The range of scores is 0 to 63, with a higher value representing a worse outcome.
Time Frame: Baseline, Months 3, 6, 9, 12, 18, 24
Population: as for outcome 29
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Standard of Care | Early Adalimumab
Number analyzed (Participants) | 33 | 38
units on a scale
  Month 3 | -4.3 (1.15) | -3.1 (1.07)
  Month 6 | -1.0 (1.28) | -2.4 (1.19)
  Month 9 | -4.3 (1.04) | -3.7 (0.97)
  Month 12 | -5.1 (1.24) | -3.5 (1.15)
  Month 18 | -4.8 (1.22) | -3.5 (1.14)
  Month 24 | -4.8 (1.15) | -3.4 (1.07)
Statistical Analysis 1: Comparison: Standard of Care vs Early Adalimumab; Month 3; Test type: Superiority or Other; p = 0.458, ANCOVA — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = 1.2, 95% CI 2-sided [-2.0 to 4.3], Standard Error of Mean 1.57
Statistical Analysis 2: Comparison: Standard of Care vs Early Adalimumab; Month 6; Test type: Superiority or Other; p = 0.419, ANCOVA — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = -1.4, 95% CI 2-sided [-4.9 to 2.1], Standard Error of Mean 1.76
Statistical Analysis 3: Comparison: Standard of Care vs Early Adalimumab; Month 9; Test type: Superiority or Other; p = 0.692, ANCOVA — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = 0.6, 95% CI 2-sided [-2.3 to 3.4], Standard Error of Mean 1.42
Statistical Analysis 4: Comparison: Standard of Care vs Early Adalimumab; Month 12; Test type: Superiority or Other; p = 0.357, ANCOVA — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = 1.6, 95% CI 2-sided [-1.8 to 5.0], Standard Error of Mean 1.69
Statistical Analysis 5: Comparison: Standard of Care vs Early Adalimumab; Month 18; Test type: Superiority or Other; p = 0.420, ANCOVA — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = 1.4, 95% CI 2-sided [-2.0 to 4.7], Standard Error of Mean 1.67
Statistical Analysis 6: Comparison: Standard of Care vs Early Adalimumab; Month 24; Test type: Superiority or Other; p = 0.380, ANCOVA — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = 1.4, 95% CI 2-sided [-1.8 to 4.5], Standard Error of Mean 1.58

31. Secondary Outcome: Likert Scale for Participant's Satisfaction With Care at Months 3, 6, 9, 12, 18 and 24
Description: Participants measured their satisfaction with care by specifying their in response to the question "How satisfied are you with the results of your RA treatment?" on a 5-point Likert scale, from the following 5 answers: not satisfied, a little satisfied, moderately satisfied, well satisfied, very well satisfied. Scores range from 1 to 5, with higher scores indicating more satisfaction with their care.
Time Frame: Months 3, 6, 9, 12, 18, 24
Population: as for outcome 29
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Standard of Care | Early Adalimumab
Number analyzed (Participants) | 35 | 38
units on a scale
  Month 3 | 3.5 (0.20) | 4.1 (0.19)
  Month 6 | 3.3 (0.19) | 4.1 (0.18)
  Month 9 | 3.7 (0.17) | 4.1 (0.17)
  Month 12 | 3.9 (0.16) | 4.2 (0.15)
  Month 18 | 4.2 (0.17) | 4.2 (0.16)
  Month 24 | 4.1 (0.16) | 4.3 (0.15)
Statistical Analysis 1: Comparison: Standard of Care vs Early Adalimumab; Month 3; Test type: Superiority or Other; p = 0.046, ANCOVA — [p-value comment as in outcome 13, analysis 1]; The a priori threshold for statistical significance is P=0.05; LS Mean Difference = 0.6, 95% CI 2-sided [0.0 to 1.1], Standard Error of Mean 0.28
Statistical Analysis 2: Comparison: Standard of Care vs Early Adalimumab; Month 6; Test type: Superiority or Other; p = 0.003, ANCOVA — [p-value comment as in outcome 13, analysis 1]; The a priori threshold for statistical significance is P=0.01; LS Mean Difference = 0.8, 95% CI 2-sided [0.3 to 1.3], Standard Error of Mean 0.27
Statistical Analysis 3: Comparison: Standard of Care vs Early Adalimumab; Month 9; Test type: Superiority or Other; p = 0.204, ANCOVA — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = 0.3, 95% CI 2-sided [-0.2 to 0.8], Standard Error of Mean 0.24
Statistical Analysis 4: Comparison: Standard of Care vs Early Adalimumab; Month 12; Test type: Superiority or Other; p = 0.227, ANCOVA — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = 0.3, 95% CI 2-sided [-0.2 to 0.7], Standard Error of Mean 0.22
Statistical Analysis 5: Comparison: Standard of Care vs Early Adalimumab; Month 18; Test type: Superiority or Other; p = 0.860, ANCOVA — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = 0.0, 95% CI 2-sided [-0.4 to 0.5], Standard Error of Mean 0.23
Statistical Analysis 6: Comparison: Standard of Care vs Early Adalimumab; Month 24; Test type: Superiority or Other; p = 0.476, ANCOVA — [p-value comment as in outcome 13, analysis 1]; LS Mean Difference = 0.2, 95% CI 2-sided [-0.3 to 0.6], Standard Error of Mean 0.22

32. Secondary Outcome: Health Care Resources Questionnaire (HCR): Medical Insurance at Baseline
Description: The HCR consists of four aspects: medical insurance, health care for RA in the past 4 weeks, hospitalization in the past 4 weeks, and out of pocket expenses incurred for the current study condition. Participants were asked whether and what type of health insurance they had. Types of Canadian insurance included: Régie de l'assurance maladie du Québec (RAMQ); Société de l'assurance automobile du Québec (SAAQ); Commission de la santé et de la sécurité du travail (CSST); Canadian Health Insurance Program (CHIP); and L'indemnisation des victimes d'actes criminals (IVAC).
Time Frame: Baseline
Population: Intent-to-treat population: all participants who were randomized, received at least one dose of study drug, and had an assessment. n=the number of participants included in the percentage calculation (n=25, 28 is the number of participants who answered that they did have health insurance).
Measure: Number; unit: percentage of participants
Arm/Group | Standard of Care | Early Adalimumab
Number analyzed (Participants) | 35 | 39
percentage of participants
  Has health insurance; n=35, 39 | 71.4 | 71.8
  1 insurance; n=35, 39 | 71.4 | 66.7
  >/= 1 insurance; n=35, 39 | 0 | 2.6
  RMAQ; n=25, 28 | 4.0 | 3.6
  SAAQ; n=25, 28 | 0 | 0
  Federal government; n=25, 28 | 0 | 3.6
  CSST; n=25, 28 | 0 | 0
  OHIP; n=25, 28 | 12.0 | 21.4
  IVAC; n=25, 28 | 0 | 0
  Blue Cross; n=25, 28 | 20.0 | 7.1
  Other; n=25, 28 | 64.0 | 64.3

33. Secondary Outcome: HCR: Medical Insurance at Final Visit
Description: as for outcome 32
Time Frame: Final Visit (up to Month 24)
Population: Intent-to-treat population: all participants who were randomized, received at least one dose of study drug, and had an assessment. n=the number of participants included in the percentage calculation (n=26, 26 is the number of participants who answered that they did have health insurance).
Measure: Number; unit: percentage of participants
Arm/Group | Standard of Care | Early Adalimumab
Number analyzed (Participants) | 33 | 37
percentage of participants
  Has health insurance; n=33, 37 | 78.8 | 70.3
  1 insurance; n=33, 37 | 78.8 | 70.3
  >/= 1 insurance; n=33, 37 | 0 | 0
  RMAQ; n=26, 26 | 0 | 3.8
  SAAQ; n=26, 26 | 0 | 0
  Federal government; n=26, 26 | 0 | 3.8
  CSST; n=26, 26 | 0 | 0
  OHIP; n=26, 26 | 11.5 | 11.5
  IVAC; n=26, 26 | 0 | 0
  Blue Cross; n=26, 26 | 11.5 | 7.7
  Other; n=26, 26 | 76.9 | 73.1

34. Secondary Outcome: HCR: Health Care for RA in the Past 4 Weeks at Baseline
Description: The HCR consists of four aspects: medical insurance, health care for RA in the past 4 weeks, hospitalization in the past 4 weeks, and out of pocket expenses incurred for the current study condition. Participants were asked about their use of health care for RA in the past 4 weeks.
Time Frame: Baseline
Population: Intent-to-treat population: all participants who were randomized, received at least one dose of study drug, and had an assessment. n=the number of participants included in the percentage calculation (n=11, 10 is the number of participants who stated that they had used healthcare for RA in the past 4 weeks).
Measure: Number; unit: percentage of participants
Arm/Group | Standard of Care | Early Adalimumab
Number analyzed (Participants) | 35 | 39
percentage of participants
  Used health care in past 4 weeks; n=35, 39 | 34.1 | 25.6
  Unscheduled visits to study doctor; n=11, 10 | 27.3 | 20.0
  Visits to another physician; n=11, 10 | 27.3 | 0
  Visits to a healthcare professional; n=11, 10 | 9.1 | 20.0
  Visit to hospital emergency room; n=11, 10 | 0 | 10.0
  Use of an ambulance service; n=11, 10 | 0 | 0
  Complementary/alternative therapy visits; n=11, 10 | 0 | 0

35. Secondary Outcome: HCR: Health Care for RA in the Past 4 Weeks at Final Visit
Description: as for outcome 34
Time Frame: Final Visit (up to Month 24)
Population: Intent-to-treat population: all participants who were randomized, received at least one dose of study drug, and had an assessment. n=the number of participants included in the percentage calculation (n=2, 3 is the number of participants who stated that they had used healthcare for RA in the past 4 weeks).
Measure: Number; unit: percentage of participants
Arm/Group | Standard of Care | Early Adalimumab
Number analyzed (Participants) | 33 | 37
percentage of participants
  Used health care in past 4 weeks; n=33, 37 | 6.1 | 8.1
  Unscheduled visits to study doctor; n=2, 3 | 0 | 0
  Visits to another physician; n=2, 3 | 0 | 33.3
  Visits to a healthcare professional; n=2, 3 | 50.0 | 33.3
  Visit to hospital emergency room; n=2, 3 | 0 | 33.3
  Use of an ambulance service; n=2, 3 | 0 | 0
  Complementary/alternative therapy visits; n=2, 3 | 0 | 0

36. Secondary Outcome: HCR: Out of Pocket Expenses Incurred for the Current Study Condition in the Past 4 Weeks at Baseline
Description: The HCR consists of four aspects: medical insurance, health care for RA in the past 4 weeks, hospitalization in the past 4 weeks, and out of pocket expenses incurred for the current study condition. Participants were asked what type of out-of-pocket expenses they had incurred for their RA in the past 4 weeks. Based on Canadian dollars.
Time Frame: Baseline
Population: Intent-to-treat population: all participants who were randomized, received at least one dose of study drug, and had an assessment. n=participants with non-zero expenses for given category, and included in the mean (SD) calculation.
Measure: Mean (Standard Deviation); unit: Canadian dollars
Arm/Group | Standard of Care | Early Adalimumab
Number analyzed (Participants) | 35 | 39
Canadian dollars
  Over-the-counter medications; n=11, 14 | 34.2 (28.1) | 60.3 (62.82)
  Health care professional payments; n=0, 2 | NA (NA) — n=0 for this arm | 60.0 (28.28)
  Medical procedures/laboratory tests; n=0, 0 | NA (NA) — n=0 for this arm | NA (NA) — n=0 for this arm
  Medical devices; n=2, 2 | 60.0 (56.57) | 97.5 (31.82)
  Healthcare or extra help at home; n=0, 1 | NA (NA) — n=0 for this arm | 80.0 (NA) — n=1 for this arm
  Transportation costs; n=17, 12 | 36.3 (19.53) | 30.3 (18.24)

37. Secondary Outcome: HCR: Out of Pocket Expenses Incurred for the Current Study Condition in the Past 4 Weeks at Final Visit
Description: as for outcome 36
Time Frame: Final Visit (up to Month 24)
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: Canadian dollars
Arm/Group | Standard of Care | Early Adalimumab
Number analyzed (Participants) | 35 | 39
Canadian dollars
  Over-the-counter medications; n=7, 7 | 108.3 (78.75) | 34.4 (32.82)
  Health care professional payments; n=1, 3 | 45.0 (NA) — n=1 for this arm | 91.7 (43.68)
  Medical procedures/laboratory tests; n=0, 0 | NA (NA) — n=0 for this arm | NA (NA) — n=0 for this arm
  Medical devices; n=0, 0 | NA (NA) — n=0 for this arm | NA (NA) — n=0 for this arm
  Healthcare or extra help at home; n=0, 0 | NA (NA) — n=0 for this arm | NA (NA) — n=0 for this arm
  Transportation costs; n=4, 4 | 61.3 (40.90) | 35.0 (17.32)

ADVERSE EVENTS:
Time Frame: Baseline through Month 24 (± 10 days) plus 70 days follow-up.
Arm/Group | Standard of Care | Early Adalimumab
Serious Adverse Events (participants affected / at risk) | 3/35 | 4/39
Other Adverse Events (participants affected / at risk) | 32/35 | 33/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard of Care (N=35) | Early Adalimumab (N=39)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 1 | 0
SURGICAL FAILURE (General disorders) | 0 | 1
HERPES ZOSTER (Infections and infestations) | 0 | 1
ACUTE MYELOID LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
LUNG NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
PSYCHOTIC DISORDER (Psychiatric disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Standard of Care (N=35) | Early Adalimumab (N=39)
ANAEMIA (Blood and lymphatic system disorders) | 3 | 1
PALPITATIONS (Cardiac disorders) | 1 | 2
DRY EYE (Eye disorders) | 3 | 0
VISION BLURRED (Eye disorders) | 2 | 1
VITREOUS FLOATERS (Eye disorders) | 2 | 1
DIARRHOEA (Gastrointestinal disorders) | 2 | 1
DYSPEPSIA (Gastrointestinal disorders) | 1 | 2
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 2 | 1
MOUTH ULCERATION (Gastrointestinal disorders) | 2 | 0
NAUSEA (Gastrointestinal disorders) | 6 | 1
VOMITING (Gastrointestinal disorders) | 2 | 0
CHEST PAIN (General disorders) | 0 | 2
CYST (General disorders) | 2 | 0
FATIGUE (General disorders) | 3 | 3
INJECTION SITE REACTION (General disorders) | 2 | 5
DRUG HYPERSENSITIVITY (Immune system disorders) | 3 | 0
CYSTITIS (Infections and infestations) | 0 | 2
HERPES ZOSTER (Infections and infestations) | 2 | 0
INFLUENZA (Infections and infestations) | 1 | 3
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 3 | 2
NASOPHARYNGITIS (Infections and infestations) | 7 | 8
ORAL CANDIDIASIS (Infections and infestations) | 0 | 2
RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 | 1
SINUSITIS (Infections and infestations) | 3 | 1
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 | 2
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 3 | 6
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 2 | 6
BLOOD CHOLESTEROL INCREASED (Investigations) | 1 | 5
BLOOD GLUCOSE INCREASED (Investigations) | 2 | 0
BLOOD TRIGLYCERIDES INCREASED (Investigations) | 3 | 3
HEPATIC ENZYME INCREASED (Investigations) | 2 | 0
WEIGHT DECREASED (Investigations) | 2 | 0
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 3 | 3
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 | 3
JOINT SWELLING (Musculoskeletal and connective tissue disorders) | 2 | 1
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 3 | 1
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 2 | 0
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 2 | 3
RHEUMATOID ARTHRITIS (Musculoskeletal and connective tissue disorders) | 8 | 10
TENDONITIS (Musculoskeletal and connective tissue disorders) | 1 | 2
AMNESIA (Nervous system disorders) | 2 | 0
DIZZINESS (Nervous system disorders) | 3 | 1
HEADACHE (Nervous system disorders) | 6 | 2
ANXIETY (Psychiatric disorders) | 2 | 2
DEPRESSION (Psychiatric disorders) | 6 | 2
INSOMNIA (Psychiatric disorders) | 2 | 1
COUGH (Respiratory, thoracic and mediastinal disorders) | 4 | 2
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 2 | 0
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 | 3
ACNE (Skin and subcutaneous tissue disorders) | 3 | 0
ALOPECIA (Skin and subcutaneous tissue disorders) | 3 | 0
DRY SKIN (Skin and subcutaneous tissue disorders) | 2 | 0
ECCHYMOSIS (Skin and subcutaneous tissue disorders) | 0 | 2
ECZEMA (Skin and subcutaneous tissue disorders) | 2 | 2
RASH (Skin and subcutaneous tissue disorders) | 5 | 4
RASH PAPULAR (Skin and subcutaneous tissue disorders) | 2 | 2
HOT FLUSH (Vascular disorders) | 0 | 2
HYPERTENSION (Vascular disorders) | 3 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.